CLINICAL TRIAL: NCT02252315
Title: Written Versus Verbal Education for Mild Traumatic Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Noah Silverberg, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H13-01647
Record Dates: First submitted 2014-08-28; First posted 2014-09-30 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

ARMS (2):
- Written Education (Active Comparator)
  Interventions: Other: Educational Brochure
- Verbal Education (Active Comparator)
  Interventions: Other: Verbal education module

INTERVENTIONS:
Other: Educational Brochure — Participants will receive written education materials about mild traumatic brain injury.
  Arms: Written Education
Other: Verbal education module — A structured in-person education module about mild traumatic brain injury.
  Arms: Verbal Education

SUMMARY:
Mild traumatic brain injury (MTBI) is a common injury that involves loss of consciousness or alteration in mental status induced by an external mechanical force to the head. Education about symptoms and reassurance of a prompt recovery usually results in full recovery. However, a subgroup appears to have persistent symptoms and disability. This study will recruit MTBI patients from two Emergency Departments with the aim of identifying modifiable patient characteristics that can delay or prevent full recovery. A secondary aim is to determine if providing education in writing or in-person makes a difference.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of a likely concussion without hospital admission
* Participants live locally with a fixed address
* Participants experience at least one new symptom

Exclusion Criteria:

* Participants who cannot understand/read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Presence of Postconcussional Syndrome | 3 Months
  The primary outcome is the presence of Postconcussion Syndrome, defined as 3+ symptoms endorsed as "mild" or greater on the Rivermead Postconcussion Symptom Questionnaire.

SECONDARY OUTCOMES:
Glasgow Outcome Scale-Extended (GOS-E) | 3 Months
  Structured interview to assess disability level.
Patient Health Questionnaire-9 (PHQ-9) | 3 Months
  Depressive symptoms questionnaire.
PTSD Checklist-Civilian version (PCL-C) | 3 Months
  Post-traumatic stress symptoms questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Silverberg, PhD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Lions Gate Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia